CLINICAL TRIAL: NCT06884410
Title: Reproducibility of Multiparametric Renal Magnetic Resonance Imaging on 1.5T MRI Scanners (RESPECT_1.5T Sub-study)
Brief Title: Reproducibility of Multiparametric Renal Magnetic Resonance Imaging on 1.5T MRI Scanners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RESPECT_1.5T
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Multiparametric MRI
Keywords: multiparametric MRI; standardization; reproducibility; kidney; MRI scanners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Healthy volunteers selected from 4 different centers. Each center will recruit 6 males and 6 females each.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Multiparametric renal MRI on 1.5T scanners

SUMMARY:
This is an interventional, multicenter, prospective study involving healthy volunteers, to primarily assess the reproducibility of multiparametric renal MRI on 1.5T scanners. The study is also aimed at assessing possible differences in renal MRI reproducibility on 1.5T MRI scanners by sex and age, and assessing possible differences in renal MRI reproducibility across field strengths (1.5T vs 3T) in the subgroup of subjects enrolled in both RESPECT clinical study and in the current subproject.

DETAILED DESCRIPTION:
Over the past decade, renal Magnetic Resonance Imaging (MRI) has emerged as a promising non-invasive technique for improved understanding and characterisation of renal pathophysiology.

Despite renal MRI potential to address several key clinical questions, current methodological differences across studies hinder reliable comparisons of the results, which can only be regarded as preliminary. Widely accepted normative values of renal MRI measures to establish benchmarks for early diagnosis, prognosis or treatment planning are not available. Standardization of acquisition and processing protocols across centres is therefore needed, and this is a necessary preliminary step towards multiparametric renal MRI wider use in clinical research and ultimate adoption in clinical practice.

The ongoing "Exploratory multicentre clinical study to assess repeatability, reproducibility, acceptability and clinical validity of multiparametric renal Magnetic Resonance Imaging (RESPECT Trial, NCT05229263)" trial will provide relevant information on repeatability and reproducibility of MRI measures obtained from multiparametric MRI scans acquired on 3T scanners, that represent the state-of-the-art for clinical research. However, 3T MRI scanners are not available in most clinical centres, where instead lower-field (1.5T) MRI scanners are much more common. Investigating reproducibility of renal MRI measures on 1.5T scanners and assessing possible differences in reproducibility across magnetic field strength would be needed towards translation of the results of the RESPECT clinical study to clinics.

The possible advantages that can derive from participating in the present research are essentially linked to the possibility to specifically assess the renal function with multiparametric MRI, that is not part of the routine clinical practice. More generally, in the long term, it will be possible for CKD patients to benefit from the results of this study that is aimed at demonstrating the reproducibility and the clinical validity of multiparametric MRI.

Participation in the study will not entail any additional risk to subjects' health. All clinical MRI safety procedures will be strictly followed. Indeed, multiparametric MRI acquisitions required by this research will be performed without the administration of contrast media and do not present risks in either short or long term.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study specific procedures
* Male and female subjects aged [18-70] years
* Office SBP values < 140 mmHg and DBP values ≤ 90 mmHg, under no antihypertensive therapy
* Normal renal function defined as: estimated glomerular filtration rate [eGFR] ≥ 60mL/min/1.73m2 (using CKD-EPI Creatinine Equation)
* Negative result upon urine testing for haematuria or proteinuria.

Exclusion Criteria:

* Previous enrollment in the present substudy
* Contraindications to MRI including caustrophobia, pregnancy, cardiac pacemakers or other MRI-incompatible prostheses
* Ongoing therapy (e.g. for diabetes, dyslipidemia, or any acute disease)
* Past or current oncological pathology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Volumes | At day 0 and from 7 to 14 days after
  Total kidney, cortical and medullary volumes (in mL)
Oxygenation | At day 0 and from 7 to 14 days after
  Renal tissue oxygenation obtained by measuring the R2* relaxation rate (in 1/ms)
Diffusion coefficient | At day 0 and from 7 to 14 days after
  Apparent diffusion coefficient (in cm2/s)
Tissue perfusion | At day 0 and from 7 to 14 days after
  Renal tissue perfusion (in mL/100mL/min)
Blood flow | At day 0 and from 7 to 14 days after
  Renal blood flow (in mL/min)
Relaxation times | At day 0 and from 7 to 14 days after
  T1 and T2 relaxation times (in ms)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, M.D., Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (4):
- Aarhus University Hospital, Aarhus, Denmark
- University Medical Center Mannheim, Medical Faculty Mannheim, Heidelberg University, Mannheim, Germany
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlinden C, Khadka J, Pesudovs K. Precision (repeatability and reproducibility) studies and sample-size calculation. J Cataract Refract Surg. 2015 Dec;41(12):2598-604. doi: 10.1016/j.jcrs.2015.06.029. No abstract available. PMID 26796439
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Selby NM, Blankestijn PJ, Boor P, Combe C, Eckardt KU, Eikefjord E, Garcia-Fernandez N, Golay X, Gordon I, Grenier N, Hockings PD, Jensen JD, Joles JA, Kalra PA, Kramer BK, Mark PB, Mendichovszky IA, Nikolic O, Odudu A, Ong ACM, Ortiz A, Pruijm M, Remuzzi G, Rorvik J, de Seigneux S, Simms RJ, Slatinska J, Summers P, Taal MW, Thoeny HC, Vallee JP, Wolf M, Caroli A, Sourbron S. Magnetic resonance imaging biomarkers for chronic kidney disease: a position paper from the European Cooperation in Science and Technology Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii4-ii14. doi: 10.1093/ndt/gfy152. PMID 30137584
- [Background] Caroli A, Pruijm M, Burnier M, Selby NM. Functional magnetic resonance imaging of the kidneys: where do we stand? The perspective of the European COST Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii1-ii3. doi: 10.1093/ndt/gfy181. No abstract available. PMID 30137582
- [Background] Xie L, Bennett KM, Liu C, Johnson GA, Zhang JL, Lee VS. MRI tools for assessment of microstructure and nephron function of the kidney. Am J Physiol Renal Physiol. 2016 Dec 1;311(6):F1109-F1124. doi: 10.1152/ajprenal.00134.2016. Epub 2016 Sep 14. PMID 27630064
- [Background] Grenier N, Merville P, Combe C. Radiologic imaging of the renal parenchyma structure and function. Nat Rev Nephrol. 2016 Jun;12(6):348-59. doi: 10.1038/nrneph.2016.44. Epub 2016 Apr 12. PMID 27067530